CLINICAL TRIAL: NCT03619109
Title: Evaluation of the Levels of C-Reactive Protein, Procalcitonin, and Lactate in a Normal Healthy Population When Tested With the Nanōmix eLab® System
Brief Title: Determination of Normal Reference Values of CRP, Procalcitonin, and Lactate Levels for the Nanōmix eLab® System
Status: Completed | Type: Observational
Sponsor: Nanomix (Industry)
Responsible Party: Sponsor
Other Study IDs: Nanomix
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2019-03-14 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: C-Reactive Protein; CRP; Procalcitonin; Lactate; In Vitro Diagnostic Product; IVD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Leftover plasma samples (without cells/ RNA/DNA) will be aliquoted and stored at Sponsor for potential future analysis/ projects.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Volunteers: No real intervention since samples from volunteers are not tested on Nanōmix eLab™ System near any volunteers. Leftover samples are stored at Sponsor for potential future analysis/ projects.

SUMMARY:
The main objective of this clinical study is to determine the normal reference range of the Nanōmix eLab® (eLab) C-Reactive Protein, Procalcitonin and Lactate Assay.

DETAILED DESCRIPTION:
The purpose of this clinical study is to determine the normal reference range of the Nanōmix eLab® (eLab) C-Reactive Protein, Procalcitonin and Lactate Assay, whereby collected blood samples are used to characterize the distribution of C-Reactive Protein (CRP), Procalcitonin (PCT), and Lactate (LAC) in a population of healthy subjects. Approximately 4 mL of whole blood will be collected by venipuncture from normal healthy volunteers and tested with the eLab C-Reactive Protein, Procalcitonin, and Lactate assay within 30 minutes of collection. Following the whole blood test, the sample will be spun down to plasma and a plasma sample will be tested on the eLab with the eLab C-Reactive Protein, Procalcitonin, and Lactate assays within 30 min of the whole blood test. Demographic and health information will also be collected from each participant by having them complete a questionnaire. The test results will be collated to establish the normal range (2.5 - 97.5th percentile) for each analyte. The remaining plasma will be frozen and stored at -80° C.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Must have provided written informed consent
* Must self-report as being in good health

Exclusion Criteria:

* Under the care of a physician and currently receiving any therapy
* Obesity (BMI > 35)
* Have had outpatient surgery or been hospitalized in the last 3 months for any reason
* Known to be pregnant or nursing
* Engaged in exertion resulting in an estimated HR>120 bpm for > 5 minutes in the last 4 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2017-12-22 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Normal reference ranges of CRP, Procalcitonin, and Lactate for the Nanōmix eLab® System | One timepoint at enrollment
  To determine the normal reference ranges of CRP, Procalcitonin, and Lactate for the Nanōmix eLab® System using Li-Heparinized venous whole blood and Li-Heparinized plasma samples from healthy subjects.System using Li-Heparinized venous whole blood and Li-Heparinized plasma samples from healthy subjects.Nanōmix eLab® System.

CONTACTS AND LOCATIONS:
Overall Officials: Tina Landess, Study Director — Nanomix
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States